CLINICAL TRIAL: NCT00783419
Title: Rate of Pelvic Inflammatory Disease and Tubo-ovarian Abscess at SMH
Brief Title: Rate of Pelvic Inflammatory Disease at St. Michael's Hospital
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 07-042
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Pelvic Inflammatory Disease
Keywords: tubo-ovarian abscess, pelvic-inflammatory disease
MeSH Terms: conditions — Pelvic Inflammatory Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A retrospective review of women who came through the ER at SMH with a pelvic inflammatory disease (PID) or tubo-ovarian abscess (TOA) between 1995-2005. They were looking at people with this diagnosis to determine how they were treated, whether as inpatient or outpatient and whether they were treated with drugs and how were these given and also did they develop an abscess.

ELIGIBILITY:
Inclusion Criteria:

* women admitted to Emergency with pelvic-inflammatory disease or tubo-ovarian abscess from the year range: 1995-2000

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with pelvic-inflammatory disease or tubo-ovarian abscess
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2007-03; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yudin, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada